CLINICAL TRIAL: NCT01673763
Title: Study to Reduce Incidence of Post-ERCP Pancreatitis by Stent Insertion in the Main Pancreatic Duct After Unintended Cannulation of the Main Pancreatic Duct
Brief Title: Post-ERCP Pancreatitis Prevention by Stent Insertion
Acronym: PEPSI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Technical University of Munich (Other)
Collaborators: Northern State University, Russia (Unknown); KU Leuven (Other); Latvijas Universitates Medicinas (Unknown)
Responsible Party: Principal Investigator, Monther Bajbouj, PD Dr. med. Hana Algül, Technical University of Munich
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 240179
Record Dates: First submitted 2011-10-17; First posted 2012-08-28 (Estimated); Last update posted 2017-10-13 (Actual); Status verified 2017-10

CONDITIONS: Post-ERCP Acute Pancreatitis
Keywords: ERCP; endoscopy; pancreatitis
MeSH Terms: conditions — Pancreatitis

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Stent (Active Comparator): Stent insertion into the main pancreatic duct
  Interventions: Device: Stent insertion into the main pancreatic duct
- No stent (No Intervention): No stent insertion into the main pancreatic duct

INTERVENTIONS:
Device: Stent insertion into the main pancreatic duct — Stent insertion into the main pancreatic duct
  Arms: Stent

SUMMARY:
The presented study is designed to analyze the efficacy of pancreatic stent insertion in patients undergoing ERCP with accidental cannulation of the pancreatic duct.

ELIGIBILITY:
Inclusion Criteria:

* all patients undergoing ERCP with unintended cannulation or opifiacation of main pancreatic duct
* age > 17 years
* signed informed consent

Exclusion Criteria:

* intention to intervene main pancreatic duct
* age < 18 years
* pregnancy
* absent of signed informed consent

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 169 (Actual)
Dates: Start 2010-07 (Actual); Primary Completion 2016-06 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Incidence of post-ERCP pancreatitis | up to 1 week

CONTACTS AND LOCATIONS:
Overall Officials: Hana Algül, MD, MPH, Principal Investigator — II. Medizinische Klinik, Klinikum rechts der Isar, Ismaniger Strasse 22, 81675 Munich
Locations (4):
- Deptartment of Hepatobiliary Diseases Leuven University Hospitals, Leuven, Belgium
- Klinikum rechts der Isar, Technische Universität München, Munich, Germany
- P. Stradin Clinical University Hospital Gastroenterology Centere Latvijas Universitates Medicinas, Riga, Latvia
- First city hospital of emergency care Northern State Medical University, Arkhangelsk, Russia